CLINICAL TRIAL: NCT00003040
Title: A Phase II Study to Evaluate Transoral CO2 Laser Supraglottic Laryngectomy and Irradiation in Stage I, II and III Squamous Cell Carcinoma of the Supraglottic Larynx
Brief Title: S9709, Laser Surgery Plus Radiation Therapy in Treating Patients With Early Stage Cancer of the Larynx
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065668; U10CA032102 (NIH); S9709 (Other: SWOG)
Record Dates: First submitted 1999-11-01; First posted 2004-03-01 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Laser Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transoral CO2 laser laryngectomy and RT (Experimental): Transoral CO2 laser supraglottic laryngectomy and irradiation
  Interventions: Procedure: laser surgery; Radiation: radiation therapy

INTERVENTIONS:
Procedure: laser surgery — CO2 supraglottic laryngectomy within 28 days following registration with neck dissection as needed
  Other Names: CO2 laser surgery
Radiation: radiation therapy — 200 cGy per day, five days per week for approximately 6 weeks, to begin 14 days after laser surgery
  Other Names: RT

SUMMARY:
RATIONALE: Laser surgery for cancer of the larynx may have fewer side effects and improve recovery. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy and laser surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of laser surgery plus radiation therapy in treating patients with early stage cancer of the larynx.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the feasibility of treating untreated stage I, II and selected stage III squamous cell carcinoma of the supraglottic larynx with endoscopic surgery and irradiation. II. Estimate the 3 year progression free survival and describe the location of disease progression.

OUTLINE: Patients receive carbon dioxide laser laryngectomy within 28 days following protocol registration. Patients with N1 disease may undergo an optional neck dissection ipsilateral to the neck mass. Neck dissection includes complete removal of at least lymph node levels 2-4. Radiation therapy begins 14 days following laser surgery. Patients are followed every 3 months for the first year, every 6 months for the second year, and every 12 months thereafter until death.

PROJECTED ACCRUAL: There will be 50 patients accrued into this study in 3 years with an estimated accrual rate of 20 patients per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, newly diagnosed, untreated stage I, II, or selected stage III (T1-T2, N1, M0) squamous cell carcinoma of the supraglottic larynx Bidimensionally measurable disease No metastatic or stage III T3 disease No immediate life-threatening complications of the disease

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: SWOG 0 or 1 Life expectancy: Not specified Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 50,000/mm3 Hemoglobin greater than 10.0 g/dL Hepatic: Not specified Renal: Not specified Cardiovascular: At least 3 months since prior myocardial infarction No uncontrolled congestive heart failure No unstable or uncontrolled angina Other: No prior malignancy except for the following: Adequately treated basal cell or squamous cell skin cancer In situ cervical cancer Other cancer for which the patient has been disease-free for at least five years No history of prior laryngeal cancer No history of primary tumors of any aerodigestive tract site except disease site All fertile patients must use an effective contraceptive method Must be medically able to undergo general anesthesia No psychological, familial, sociological or geographical conditions that do not permit medical follow-up and compliance with study protocol No other unstable or pre-existing major medical condition

PRIOR CONCURRENT THERAPY: No prior treatment for squamous cell carcinoma of the supraglottic larynx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1997-09; Primary Completion 2007-02 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
feasibility | 4 years
  To test the ability to accrue patients to the study at a rate compatible with efficiency (20 patients per year).

SECONDARY OUTCOMES:
progression-free survival | 3 years
  From date of registration to date of first observation of progressive disease, death due to any cause or early discontinuation of treatment
return to swallowing function | two weeks
  how long patients require feeding tubes and the proportion of patients requiring tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Roy K. Davis, MD, Study Chair — University of Utah
Locations (12):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Oregon Cancer Center, Portland, Oregon
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Result] Agrawal A, Moon J, Davis RK, Sakr WA, Giri SP, Valentino J, LeBlanc M, Truelson JM, Yoo GH, Ensley JF, Schuller DE; Southwest Oncology Group. Transoral carbon dioxide laser supraglottic laryngectomy and irradiation in stage I, II, and III squamous cell carcinoma of the supraglottic larynx: report of Southwest Oncology Group Phase 2 Trial S9709. Arch Otolaryngol Head Neck Surg. 2007 Oct;133(10):1044-50. doi: 10.1001/archotol.133.10.1044. PMID 17938330